CLINICAL TRIAL: NCT03608540
Title: A Prospective Study to Evaluate the Safety and Feasibility of an Endoluminal-suturing Device (Endomina TM) as an Aid for Endoscopic Full Thickness Resection
Brief Title: Endomina as an Aid for Endoscopic Full Thickness Resection
Acronym: EFTR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrolment too slow
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2018/263
Record Dates: First submitted 2018-07-10; First posted 2018-08-01 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Submucosal Tumor of Intestine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Suturing system with suture apposition then bulging formation then cutting the lesion
  Interventions: Device: Endomina

INTERVENTIONS:
Device: Endomina — Suturing system with sutures apposition then bulging then cutting

SUMMARY:
The concept of natural orifice transluminal endoscopic surgery (NOTES) (1) has evolved to endoscopic full thickness resection (EFTR). It represents innovation in technique that allows endoscopists to advance further into the endoscopic surgical space. EFTR has transformed the ability to tackle subepithelial tumors (SETs) and early mucosal neoplasm that are not amenable to classic ESD technique, enhance the staging accuracies for marginal lesions, and even increase the diagnostic capabilities for infiltrative disorders. Thus far, multiple methods have been described to perform EFTR, including nonexposed and exposed techniques, with the closure occuring before resection or after resection, respectively (2). Early comparative studies show no difference between the two methods (3). However, the procedures themselves are limited by the current tools available and by described techniques to achieve resection.

Investigators are described here a novel non-exposed technique, with closure before resection, using the Endomina device.

ELIGIBILITY:
Inclusion Criteria:

1. Lesion untreatable with standard technique.
2. Age between 18-65 years;
3. Must be able to comply with all study requirements for the duration of the study as outlined in the protocol. This includes complying with the visit schedule as well as study specific procedures such as: clinical assessment, endoscopy, radiography, as well as laboratory investigations;
4. Must be able to understand and be willing to provide written informed consent;
5. Must live within 75 km of the treatment site;

Exclusion Criteria:

1. Achalasia and any other esophageal motility disorders (for upper GI lesion)
2. Severe esophagitis (for upper GI lesion)
3. Gastro-duodenal ulcer (for upper GI lesion)
4. Severe renal, hepatic, pulmonary disease or cancer;
5. GI stenosis or obstruction;
6. Pregnancy, breastfeeding or willing to become pregnant in the coming 18 months;
7. Anticoagulant therapy;
8. Impending gastric surgery 60 days post intervention (Upper GI);
9. Currently participating in other study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Incidence of all Adverse Device Effects | one year from procedure
  Safety will be characterized by the incidence of all Adverse Device Effects

SECONDARY OUTCOMES:
R0 resection | 1 month after resection
  R0 resection at histology

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Department Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No